CLINICAL TRIAL: NCT01343030
Title: Prospective Radiologic Evaluation of Changes That Might Affect Breast Cancer Diagnosis Following Fat Grafting and Silicone Breast Implants
Brief Title: Prospective Radiologic Evaluation of Changes Following Fat Grafting
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: The Institute for Basic and Applied Research in Surgery (Unknown); Mentor Worldwide, LLC (Industry); Clinique SPONTINI (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1011M93112; IBARS (Other Grant/Funding Number: G10-0068)
Record Dates: First submitted 2011-03-22; First posted 2011-04-27 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with implants: Patients with silicone implants and fat grafting.

SUMMARY:
Breast implants are currently used for cosmetic breast augmentation and in breast reconstruction following mastectomy for breast cancer. Fat grafting is a technique where fat is injected around the periphery of a breast implant to camouflage the transition between implant and the body. The investigators propose to show mammography images of women who have had breast implants with fat grafting to informed and blinded radiologists and evaluate their readings of the images.

Hypothesis: with mammographic screening, radiologists will be able to distinguish between findings associated with fat grafting and those which are suspicious for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women with silicone implants and fat grafting

Exclusion Criteria:

* Procedures performed outside the University of Minnesota or Clinique Spontini Paris, France

Ages: 18 Years to 84 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will select patients from Clinique Spontini Paris France and from patients at the University of Minnesota USA who have undergone placement of silicone breast implants with fat grafting.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Radiologist dictations of mammograms | We will obtain mammograms and MRIs of participants at intervals of 6 months for up to 24 months post fat grafting.
  We will compare the Bi-Rad level score readings, and recommended follow-up of the blinded and non-blinded radiologist's read of study participants mammograms.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce L Cunningham, MD, Principal Investigator — University of Minnesota
Locations (2):
- University of Minnesota, Minneapolis, Minnesota, United States
- Clinique SPONTINI, Paris, France